CLINICAL TRIAL: NCT01543971
Title: Phase I Double-Blinded Comparison Study Using TXA127 and/or Neupogen to Increase Peripheral Blood Stem Cell (CD34+) Counts
Brief Title: Safety and Efficacy of TXA127 and Neupogen to Increase Peripheral Blood Stem Cells (PBSCs)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tarix Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TXA127-2009-003
Record Dates: First submitted 2010-02-10; First posted 2012-03-05 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Miscellaneous Peripheral Blood Cell Abnormalities
Keywords: Peripheral blood stem cell mobilization; CD34+ count
MeSH Terms: interventions — angiotensin I (1-7); Filgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TXA127 (Active Comparator): (Group A) TXA127 at 300 mcg/kg once a day for 5 days
  Interventions: Drug: TXA127
- Neupogen (Active Comparator): (Group B) Neupogen 10 mcg/kg once a day for 5 days
  Interventions: Drug: Neupogen (filgrastim)
- TXA127 and Neupogen (Active Comparator): (Group C) both TXA127 (300mcg/kg) and Neupogen (10mcg/kg) together once a day for 5 days
  Interventions: Drug: TXA127; Drug: Neupogen (filgrastim)

INTERVENTIONS:
Drug: TXA127 — TXA127 : 300mcg/kg per day for 5 days, injection
  Other Names: filgrastim; angiotensin 1-7
  Arms: TXA127; TXA127 and Neupogen
Drug: Neupogen (filgrastim) — Neupogen : 10mcg/kg per day for 5 days, injection
  Other Names: filgrastim; angiotensin 1-7
  Arms: Neupogen; TXA127 and Neupogen

SUMMARY:
This is a Phase I Study to be conducted in 18 healthy volunteers. Each will receive daily injections for 5 days of TXA127 alone, or Neupogen alone, or TXA127 plus Neupogen together.

The aim of the study is to determine the safety of the TXA127 alone and in combination with Neupogen, and to determine whether the use of TXA127 alone or in combination with Neupogen enhances peripheral blood stem cell (CD34+)mobilization.

DETAILED DESCRIPTION:
In this double-blinded comparison study, healthy volunteers will be randomized to one of 3 treatment groups: (Group A) TXA127 at 300 mcg/kg once a day for 5 days or (Group B) Neupogen 10 mcg/kg once a day for 5 days or (Group C) both together once a day for 5 days, these treatments administered by subcutaneous injection, to increase peripheral blood stem cell (CD34+) concentrations in healthy volunteers.

A minimum of 18 healthy male and female volunteer Subjects (6 in each treatment group) who meet all inclusion and none of the exclusion criteria will be enrolled in this study. Subjects will be recruited from the study center's existing database of healthy volunteers and/or by advertising. A sufficient number of alternate volunteers will be screened and checked-in on Day 0 to ensure 6 eligible healthy volunteers are enrolled on Day 1 in each treatment group. Subjects will remain housed in teh Unit during the conduct of this study.

Safety: Predose blood samples will be collected immediately prior to receiving the study medication(s), as well as at 4 hours, 8 hours, 12 hours and 16 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer is capable of reading, understanding and complying with the protocol, has been informed of the nature and risks of study participation and has signed the informed consent document prior to undergoing any study related procedures.
* Volunteer is male or female and is 18 to 45 years of age, inclusive. If female, must be non-lactating and have a negative serum pregnancy test result at screening and on admission.
* Must be in good health and must weigh at least 45 kg, but not more than 90 kg and have a Body Mass Index (BMI) between 17.5 kg/m2 and 35 kg/m2.
* Screening and admission clinical laboratory test results that are within lab's reference range or, if not, are considered not clinically significant by the Investigator.
* Screening and admission 12-lead electrocardiograms (ECGs) that are normal or, if abnormal, are considered not clinically significant by the Investigator.
* Have negative urine drug and alcohol toxicology screens at screening and on admission, with negative HIV antibody and hepatitis panel results at screening.

Exclusion Criteria:

* History of acute or chronic medical condition or test abnormality that would significantly increase Volunteer's risk of study participation or significantly increase risk of not achieving study objectives, in the Investigator's opinion.
* Has known or suspected liver disease (active hepatitis, cirrhosis, hepatic insufficiency or ascites) or has a transaminase value > 2x ULN or total bilirubin > 1.5 x ULN, a history of spleen enlargement, except if due to infectious mononucleosis resolved more than 6 months prior to scheduled admission, or a current finding of spleen enlargement. Has a history of mononucleosis within previous six months of scheduled admission.
* Has an abnormally low Protein C or Protein S at screening, or screening laboratory tests indicate Factor V Leiden is present.
* Has a history of venous thrombosis or pulmonary embolism, or has systolic blood pressure persistently >145 mm Hg or <90 mm Hg, or diastolic blood pressure persistently >90 mm Hg or <60 mm Hg at screening or on admission.
* Has a heart rate persistently >90 beats/minute or <45 beats/minute on vital signs testing at screening or on admission, or a 10-second ECG at Screening, Admission or Baseline (prior to first dose) showing any of the following:

  * HR that is < 45 or > 90 bpm;
  * QRS interval that is > 120 msec;
  * PR interval that is <120 or >220 msec;
  * QTcF that is < 300 msec or > 450 msec;
  * Any fascicular block or bundle branch block;
  * Neuromuscular ECG artifact that cannot be readily eliminated.
* Has a history of substance abuse, drug addiction, or alcoholism within 1 year prior to screening. (As defined by DSM IV criteria).
* Within 2 weeks prior to scheduled administration of study drug, Volunteer has taken any prescription or over-the-counter medication, herbal preparation or dietary supplement that, in the opinion of the Investigator, may increase risk to Volunteer's safety or to achievement of study objectives.
* Unwilling to abstain from alcohol use or from caffeine from 24 hours prior to admission.
* Has donated blood or blood products within 30 days prior to admission; is considered mentally unstable or exhibits anxious, excitable, hostile, or emotionally reactive affect; has received an investigational test substance within 30 days prior to the scheduled administration of investigational test article, or anticipates receiving any investigational test substance other than TXA127 during the course of this study.
* Volunteer has previously participated in a clinical study of TXA127.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-12; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Assessed daily during dosing (Days 1 - 5) and at the two follow up visits (Day 7 and Day 12).
  In this phase I study the primary safety variables being assessd include laboratory variables (chemistry, hematology, coagulation system parameters, and urinalysis) and regular vital signs, injection site inspection, and physical exams as indicated.

SECONDARY OUTCOMES:
Preliminary effectiveness as assessed by changes in the concentration of peripheral blood stem cells (CD34+) and other hematologic parameters. | Daily assessment during dosing (Days 1 - 5) and at the two follow up visits (Days 7 and 12)
  Parameters being assessed for preliminary effectiveness in this phase I study include routine chemistry and hematology parameters and flow-cytometric evaluation of blood samples for CD34, CD3, CD4, CD8 and CD19 concentrations at 4, 8, 12 and 16 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Gere diZerega, MD, Study Director — US Biotest, Inc.
Locations (1):
- Charles River Clinical Servies Norhtwest, Tacoma, Washington, United States